CLINICAL TRIAL: NCT07310641
Title: Descriptive Analysis of Couples With Polycystic Kidney Disease (PKD) Accessing the Arco Hospital Assisted Reproductive Technology Center for Preimplantation Testing and Comparing Outcomes and Complications in Autosomal Dominant Polycystic Kidney Disease (ADPKD) Couples in Which the Male is a Carrier of the Disease Versus Couples in Which the Female is a Carrier
Brief Title: Descriptive Analysis of Preimplantation Genetic Test (PGT)in Couples With Polycystic Kidney Disease (PKD). In the ADPKD Subgroup Evaluation of Outcomes and Complications Comparing Couples in Which the Father is Affected With Couples in Which the Mother is Affected
Acronym: PGT-M PKD
Status: Completed | Type: Observational
Sponsor: Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other)
Responsible Party: Sponsor
Other Study IDs: 28258
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Kidney Disease; Assisted Reproductive Technology; Preimplantation Genetic Testing (PGT)
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with autosomal dominant polycystic kidney disease
  Interventions: Procedure: Assisted reproductive technology and preimplantation diagnosis for monogenic diseases
- Subjects with autosomal recessive polycystic kidney disease
  Interventions: Procedure: Assisted reproductive technology and preimplantation diagnosis for monogenic diseases

INTERVENTIONS:
Procedure: Assisted reproductive technology and preimplantation diagnosis for monogenic diseases — Assisted reproductive technology and preimplantation diagnosis for monogenic diseases

SUMMARY:
The goal of this observational study is to evaluate the outcomes of assisted reproductive technology (ART) combined with preimplantation genetic testing for monogenic diseases (PGT-M) in couples affected by or carriers of polycystic kidney disease (PKD). The participant population includes couples in which one partner has autosomal dominant polycystic kidney disease (ADPKD) or both partners have autosomal recessive polycystic kidney disease (ARPKD), who were treated at the Arco Medically Assisted Procreation Center (part of Azienda Provinciale per i Servizi Sanitari della Provincia Autonoma di Trento) between January 1, 2018, and August 1, 2024, and who provided informed consent to participate in the study.

The main questions it aims to answer were:

* What are the outcomes in terms of clinical pregnancy and live birth rates in this population undergoing ART with PGT-M?
* What is the incidence of complications, including ovarian hyperstimulation syndrome (OHSS), miscarriage, hypertension, and preeclampsia, in these patients?

There is no external comparison group; however, the study may perform internal comparisons between subgroups (e.g., ADPKD vs ARPKD couples) to assess whether specific forms of PKD are associated with different reproductive outcomes.

Participants have:

1. Undergone ART procedures including ovarian stimulation, oocyte retrieval, fertilization, embryo biopsy, and transfer of embryos free of the pathogenic mutation.
2. Received genetic counseling and preimplantation genetic testing for monogenic diseases (PGT-M).
3. Been monitored throughout the process for clinical outcomes and complications (e.g., OHSS, pregnancy loss, hypertensive disorders).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Member of a heterosexual couple in which one of the two individuals is affected by ADPKD (with the condition confirmed by genetic diagnosis), or in which both members are carriers of ARPKD (with the condition genetically confirmed), who have been taken in charge by the Arco Medically Assisted Procreation (MAP) Center between January 1, 2018, and August 1, 2024, for the purpose of preimplantation genetic testing for monogenic diseases (PGT-M).
* Couples in which both partners have given their consent to participate in the study and to the processing of personal data.

Exclusion Criteria:

* Minors
* Couples in which one or both members have not given their consent to participate in the study and to the processing of personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Couples carrying polycystic kidney disease referred to the ART center at Arco Hospital, seeking to undergo preimplantation genetic testing and achieve a pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Live birth or ongoing pregnancy at term during the observation period | From January 2018 to July 2024

SECONDARY OUTCOMES:
Live birth - ongoing pregnancy | From January 2018 to July 2024
Number and percentage of preterm births (<37 weeks) in each cohort | From January 2018 to July 2024
Incidence of pregnancy complications in the two cohorts | From January 2018 to July 2024
Number of miscarriages in each cohort | From January 2018 to July 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Arco, Arco, Trento, Italy